CLINICAL TRIAL: NCT01343823
Title: Evaluation of Ecallantide for the Acute Treatment of Angiotensin Converting Enzyme Inhibitor Induced Angioedema
Brief Title: Evaluation of Ecallantide for Treatment of Angiotensin Converting Enzyme (ACE) Inhibitor Induced Angioedema
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim analysis suggested a trend favoring ecallantide; observed response rate to placebo was substantially higher than described in medical literature.
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DX-88/27
Record Dates: First submitted 2011-04-27; First posted 2011-04-28 (Estimated); Results first posted 2013-11-18 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-05

CONDITIONS: ACE Inhibitor Induced Angioedema
MeSH Terms: interventions — ecallantide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ecallantide 10mg (Active Comparator): Administered as one 3 mL SC injection containing 10 mg ecallantide and one 3 mL SC injection of matching placebo.
  Interventions: Drug: ecallantide 10 mg; Drug: placebo match for 10 mg ecallantide arm
- placebo (Placebo Comparator): Administered as two SC 3 mL injections
  Interventions: Drug: placebo
- ecallantide 60mg (Active Comparator): Administered as two 3 mL SC injections, each containing 30 mg ecallantide
  Interventions: Drug: ecallantide 60 mg
- ecallantide 30mg (Active Comparator): Administered as one 3 mL SC injection containing 30 mg ecallantide and one 3 mL SC injection of matching placebo.
  Interventions: Drug: ecallantide 30 mg; Drug: placebo match for 30 mg ecallantide arm

INTERVENTIONS:
Drug: ecallantide 60 mg — Administered as two 3 mL SC injections, each containing 30 mg ecallantide
  Arms: ecallantide 60mg
Drug: ecallantide 30 mg — Administered as one 3 mL SC injection containing 30 mg ecallantide
  Arms: ecallantide 30mg
Drug: ecallantide 10 mg — Administered as one 3 mL SC injection containing 10 mg ecallantide.
  Arms: ecallantide 10mg
Drug: placebo — Administered as two SC 3 mL injections
  Arms: placebo
Drug: placebo match for 30 mg ecallantide arm — One 3 mL SC injection of matching placebo given to subjects randomized to the 30 mg ecallantide arm.
  Arms: ecallantide 30mg
Drug: placebo match for 10 mg ecallantide arm — One 3 mL SC injection of matching placebo given to subjects randomized to the 10 mg ecallantide arm.
  Arms: ecallantide 10mg

SUMMARY:
A double-blind, randomized, controlled trial comparing the safety and effectiveness of conventional therapy with ecallantide to conventional therapy with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 years of age or older
* Must currently be on ACE inhibitor therapy and have received a dose within 36 hours
* Presenting with ACEIA of the head/neck region within 12 hours after onset
* All females must have a negative urine pregnancy test prior to administration of the study drug. Those who have had a total hysterectomy, bilateral oophorectomy or are two years post-menopausal do not require a pregnancy test.

Exclusion Criteria:

* Hypersensitivity to ecallantide
* Pregnancy or breast feeding
* Patients who have had angioedema and were not concurrently on an ACE inhibitor
* Patients exhibiting urticaria
* Patients who are intubated or who have a tracheostomy related to the current episode of angioedema
* Opinion of the investigator that the patient would not be a good candidate
* Participation in another investigational study within 30 days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2011-06-01 (Actual); Primary Completion 2012-06-01 (Actual); Study Completion 2012-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (39):
- United States (39):
  - Er Med, Llc, Montgomery, Alabama
  - Arrowhead Regional Medical Center, Colton, California
  - University of California Los Angeles School of Medicine, Los Angeles, California
  - University of California San Diego Mecial Center, San Diego, California
  - Christiana Hospital, Department of Emergency Medicine, Newark, Delaware
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Tampa General Hospital, Tampa, Florida
  - Georgia Health Sciences University, Augusta, Georgia
  - DeKalb Medical, Decatur, Georgia
  - University Consultants in Allergy and Immunology, Chicago, Illinois
  - Mercy Hospital and Medical Center, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Henry Ford Hospital, Detroit, Michigan
  - Beaumont Hospital, Royal Oak, Royal Oak, Michigan
  - Beaumont Hospital, Troy, Troy, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Nevada Acess to Research and Education Study, Las Vegas, Nevada
  - Kings County Hospital Center, Brooklyn, New York
  - Winthrop University Hospital, Mineola, New York
  - Staten Island University Hospital, Staten Island, New York
  - East Carolina University, Greenville, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - The MetroHealth System, Cleveland, Ohio
  - University Hospital East, Columbus, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University Medical Center Brackenridge, Austin, Texas
  - St Joseph Regional Health Center, Bryan, Texas
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - Emergency Medicine Residency Program, Fort Worth, Texas
  - 301 University Blvd., Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia

REFERENCES:
- [Result] Lewis LM, Graffeo C, Crosley P, Klausner HA, Clark CL, Frank A, Miner J, Iarrobino R, Chyung Y. Ecallantide for the acute treatment of angiotensin-converting enzyme inhibitor-induced angioedema: a multicenter, randomized, controlled trial. Ann Emerg Med. 2015 Feb;65(2):204-13. doi: 10.1016/j.annemergmed.2014.07.014. Epub 2014 Aug 30. PMID 25182544

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Administered by two subcutaneous injections.
- Ecallantide 10 mg: 10 mg administered as one 10 mg SC injection of ecallantide and one matching placebo
- Ecallantide 30 mg: 30 mg administered as one 30 mg SC injection of ecallantide and one matching placebo
- Ecallantide 60mg: 60 mg administered as two 30 mg SC injections of ecallantide
Period: Overall Study
Arm/Group | Placebo | Ecallantide 10 mg | Ecallantide 30 mg | Ecallantide 60mg
Started | 20 | 20 | 19 | 20
Completed | 18 | 20 | 19 | 19
Not Completed | 2 | 0 | 0 | 1
Not completed — Study Terminated | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 2 patients did not complete because the study terminated early and one patient did not complete because they withdrew from the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ecallantide 10 mg | Ecallantide 30 mg | Ecallantide 60 mg | Placebo | Total
Number analyzed (Participants) | 20 | 19 | 19 | 18 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 14 | 13 | 12 | 54
  >=65 years | 5 | 5 | 6 | 6 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 8 | 9 | 11 | 41
  Male | 7 | 11 | 10 | 7 | 35
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 19 | 19 | 18 | 76

OUTCOME MEASURES:

1. Primary Outcome: Safety and Efficacy of Ecallantide
Description: Compare the proportion of patients meeting prespecified discharge criteria in the group receiving ecallantide with conventional therapy to patients receiving placebo with conventional therapy. Patients were evaluated against 6 discharge eligibility criteria at 1,2,3,4,5, and 6 hours after study drug administration or until discharged from the ER. A responder was defined as a patient meeting all six discharge eligibility criteria as below: • Improvement of edema to "a little better" or "a lot better" as assessed by health care provider using a five point scale • Stable vital signs (within an acceptable range) • Absence of stridor • Absence of dyspnea or use of accessory muscles during respiration • Absence of drooling • Able to drink without difficulty
Time Frame: 6 hours
Population: Safety Population
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Placebo | Ecallantide 10 mg | Ecallantide 30 mg | Ecallantide 60 mg
Number analyzed (Participants) | 18 | 20 | 19 | 19
participants | 13 [NA to NA] — Not calculated | 17 [-18.8 to 43.1] | 17 [-15.9 to 45.9] | 17 [-15.9 to 45.9]

2. Secondary Outcome: Time to Symptom Resolution Based on the Visual Analog Scale (VAS)
Description: Compare the time to onset of symptom resolution between the ecallantide-treated and placebo-treated groups. The patient assessed severity of the angioedema attack using a VAS at baseline and following study drug administration every 15 minutes for the first 2 hours and then every 30 minutes through 6 hours post dosing or until the time of discharge from the ER (whichever occurred first). The scale ranged from "totally resolved" to "very severe".
Time Frame: 6 hours
Population: Time to Symptom Resolution Based on the VAS (Safety Population)
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Placebo | Ecallantide 10 mg | Ecallantide 30 mg | Ecallantide 60 mg
Number analyzed (Participants) | 18 | 20 | 19 | 19
hours | 0.50 [0.25 to 1.50] | 0.30 [0.25 to 0.73] | 0.27 [0.23 to 1.00] | 0.50 [0.22 to 2.02]

ADVERSE EVENTS:
Arm/Group | Ecallantide 10 mg | Ecallantide 30 mg | Ecallantide 60 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 6/20 | 8/19 | 8/19 | 5/18
Other Adverse Events (participants affected / at risk) | 7/20 | 11/19 | 12/19 | 8/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ecallantide 10 mg (N=20) | Ecallantide 30 mg (N=19) | Ecallantide 60 mg (N=19) | Placebo (N=18)
Angioedema (Skin and subcutaneous tissue disorders) | 5 (19) | 6 | 7 | 4
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
ECG T Wave Abnormal (Investigations) | 1 (1) | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 (1) | 0 | 0 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 (1) | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Angioedema (Epiglottic) (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Angioedema (Laryngeal) (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Carotid Artery Stenosis (Nervous system disorders) | 0 | 0 | 1 | 0
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ecallantide 10 mg (N=20) | Ecallantide 30 mg (N=19) | Ecallantide 60 mg (N=19) | Placebo (N=18)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 2
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
GERD (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0
Injection Site Pain (General disorders) | 0 | 0 | 1 | 0
Injection Site Swelling (General disorders) | 1 | 0 | 0 | 0
Gastrointestinal Viral Infection (Infections and infestations) | 1 | 0 | 0 | 0
Oral Candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
aPTT Prolonged (Investigations) | 0 | 0 | 1 | 0
Blood Alkaline Phosphatase Increase (Investigations) | 0 | 0 | 1 | 0
Blood Creatinine Increase (Investigations) | 0 | 1 | 0 | 0
Blood Glucose (Investigations) | 0 | 0 | 0 | 1
Blood Potassium Abnormal (Investigations) | 0 | 0 | 0 | 1
ECG T Wave Abnormal (Investigations) | 1 | 0 | 0 | 0
GGT Increase (Investigations) | 0 | 0 | 1 | 0
Platelet Count Decrease (Investigations) | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Carotid Artery Stenosis (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 0 | 0 | 0
Allergic Respiratory Symptom (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oopharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 5 | 8 | 7 | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The study was determined to be inadequately powered to detect a statistically significant difference between ecallantide and placebo for the primary efficacy endpoint, and therefore terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Dyax agreements vary, but Dyax will not prohibit any investigator from publishing. Dyax reviews publications prior to public release and can request deferral by up to 60 days beyond the proposed publication date if necessary to preserve its intellectual property. Dyax can request changes to publications to remove non-study-related confidential information. Dyax can also request deferral of single-center publications until after disclosure of the clinical trial's primary publication.